CLINICAL TRIAL: NCT05927623
Title: Multifaceted Intervention Using Telehealth to Reduce the Risk of Falls and Fractures in Older Men (MisterFit): A Pilot Study
Brief Title: Multifaceted Intervention Using Telehealth to Reduce the Risk of Falls and Fractures in Older Men
Acronym: MisterFIt
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Suzanne Morin, Dr., McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-37-2022-8396
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Osteoporosis; Osteoporotic Fractures; Osteoporosis, Age-Related; Muscle Loss; Men; Aging
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures; Muscular Atrophy; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Assessor-blind parallel group multicenter pilot RCT of 12 months duration.
Who Masked: Outcomes Assessor
Masking Description: Physical measures including balance, muscle strength, and gait speed will be recorded by an outcome assessor blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misterfit online group (Experimental): The Misterfit online group will receive a 12-month virtually-delivered fracture prevention intervention that includes a personalized gender-tailored strength training and balance-based exercise program, nutritional counselling and fall and fracture prevention education.
  Interventions: Behavioral: Multifaceted Virtual Fracture Prevention Program
- MisterFit offline group (Other): The Misterfit offline group will act as an attention control group receiving a fracture prevention intervention with the same components as the experimental group, but the components will not be virtual, personalized or gender-tailored.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Multifaceted Virtual Fracture Prevention Program — * Personalized exercise prescription: Comprised of muscle strengthening and balance exercises to perform three times a week, delivered and monitored remotely via the MisterFit app, a branded version of the secure commercially available Wibbi app (wibbi.com) and monthly virtual exercise consultations.
  * Virtual nutrition counseling from a registered dietitian in months 2, 4 and 6: to encourage participants to meet daily targets for calcium and vitamin D (preferably from diet), and protein intake to support muscle accretion and target weight maintenance
  * Virtual interactive information sessions in month 4 and 8: to education participants on topics identified as important by the Misterfit patient partner advisory committee.
  Arms: Misterfit online group
Behavioral: Attention Control — * Encouraged to meet the 24-Hour Movement Guidelines for adults aged 65 years or older (https://csepguidelines.ca) with telephone contacts at the same frequency that the Misterfit online group receives virtual exercise consultations
  * Nutritional fact sheets: sent by e-mail at the same frequency that the Misterfit online group meets with the research dietitian.
  * Educational fact sheets: sent by e-mail at the same frequency that the Misterfit Online group has virtual interactive information sessions
  Arms: MisterFit offline group

SUMMARY:
Men sustain over one-third of osteoporosis-related fractures worldwide. The burden of osteoporotic fractures in older men is substantial, and men suffer significantly worse fracture-related outcomes than women. Following a fracture, men sustain greater rates of subsequent fractures, loss of autonomy, and mortality than women and the imminent risk of re-fracture is several times higher in men than in women. Functional mobility, known to predict falls and fractures, is also notably worse in men following a fracture. In the fiscal year 2007-08, the overall annual costs of osteoporosis in Canadian men was evaluated to be $910 million.

Osteoporosis is primarily considered a disease of older women, and men are remarkably under-evaluated and under-treated for it. Recognition of sex and gender influences on skeletal health in men has been very slow; akin to the gap in cardiovascular diseases, where women are far less likely to receive guideline-recommended investigations and treatment.

Over 85% of Canadian men who suffer from fragility fractures do not receive osteoporosis screening and/or treatment strategies. The existence of this care gap in men underscores our current struggle to overcome important barriers including: 1) men's lack of awareness of the critical impact of osteoporosis and fractures on several aspects of their lives, and of the benefits of treatment; and 2) the absence of comprehensive and accessible treatments tailored to men.

Informed by the Knowledge-to-Action framework, we aim to address these barriers by adapting interventions with proven efficacy to engage men at high fracture risk in health behaviour change.

The current protocol is for a pilot RCT to determine the feasibility of recruitment and retention, adherence to, and acceptability of the virtually-delivered fracture prevention intervention only.

Our long-term goal is to conduct a large pragmatic randomized controlled trial (RCT) to address the research question: In older adults at high risk for fractures who self-identify as men, does anti-osteoporosis pharmacotherapy in conjunction with a virtually-delivered intervention that includes a gender-tailored strength training and balance based exercise program and nutritional counselling, improve functional mobility compared to anti-osteoporosis pharmacotherapy in conjunction with an attention control intervention.

DETAILED DESCRIPTION:
The current proposal for this assessor-blind parallel group multicenter pilot RCT of 12 months duration is in line with published frameworks for pilot studies in preparation for RCTs. For the pilot study, the investigators will enroll participants irrespective of anti-osteoporosis medication use.

This pilot RCT will determine the following primary feasibility objectives which will be assessed at 12 months :

1. Study recruitment rates: The study will be considered feasible if the investigators can recruit 12 participants per site within one year. Recruitment of 12 participants/site/year will translate to 360 participants with 10 sites over 3 years, which is the estimated sample size required for our future RCT with primary outcomes of physical function and fall rates, and secondary outcomes of bone strength.
2. Study retention rates: The study will be considered feasible if ≥ 75 % of the sample completes the 12-month assessment. This estimation is based on exercise RCTs where the attrition rate at 12 months ranged between 4% to 13% in community-based healthy men and up to 17% in frail older men.
3. Adherence to the exercise and nutrition interventions: The exercise intervention will be considered feasible if participants complete ≥ 65% of the prescribed number of exercise sessions at the 12-month follow-up. Beneficial effects of in-person supervised exercise on physical function in older men and women have been shown with a mean exercise session adherence of 60% at 12 months, and with a mean exercise session adherence of 63% in older men at 18 months. The nutrition intervention will be considered feasible if participants attend 66% of the visits.
4. Perceived usability of the telehealth platform application: via the System Usability Scale (SUS) where scores range from 0 (very poor) to 100 (excellent). Usability will be deemed to be acceptable if the mean SUS score is above 68 (SUS ≥ 68 = average user experience).

The investigators will also report exploratory analyses comparing the effect of the virtual intervention group to an attention control group. Exploratory outcomes will include the number of falls and fractures, changes in physical function (measured by lower extremity strength, gait speed, and balance), fall self-efficacy, quality of life and self-management behaviors in nutrition and exercise.

ELIGIBILITY:
Community-dwelling individuals ≥ 60 years who self-identify as men will be considered eligible if their risk for fracture is evaluated to be high, defined by the presence of one of the following inclusion criteria:

* Individuals on a Heath Canada-approved anti-osteoporosis medication (oral or intravenous bisphosphonate, denosumab, teriparatide, or romozosumab) to reduce fracture risk
* Prior hip or clinically diagnosed vertebral fracture or prior multiple fragility fractures since age 40
* Fracture at any skeletal site (excluding skull, hands, and feet) within the previous 2 years
* Ten-year probability of major osteoporotic fracture of ≥20% using the FRAX tool
* BMD T-score of ≤ -2.0 (performed as part of usual clinical care) WITH either the presence of one or more moderate or severe vertebral fractures on spine radiography OR the presence of ≥1 comorbidities (Diabetes Type I or Type II if on treatment, Parkinson's disease, congestive heart failure, chronic obstructive pulmonary disease (COPD) with previous systemic corticosteroid exposure, prostate cancer with current or prior recent (≤ 2 years) use of hormonal therapy) OR ≥ 2 falls in the previous year
* BMD T-score of ≤ -2.5 and ≥ 70 years of age

Exclusion Criteria:

* Inability to communicate in English or French;
* No access to a mobile device, tablet, or computer with a camera;
* Clinical or symptomatic spine fracture in the last 4 months, or a lower/upper limb fracture in the last 2 months;
* Uncontrolled medical comorbidity including but not limited to congestive heart failure exacerbation in the last 12 months or COPD exacerbation in the last 3 months
* Currently doing or planning to start doing either: A) Resistance training exercises with a self-rated intensity of very hard (e.g., rated ≥ 8 on a scale from 0-10) for two or more times a week OR B) Exercises to improve balance for two or more times a week
* Unable to perform basic activities of daily living or severe cognitive impairment or terminal illness
* Presence of absolute exercise contraindications unless physician approval is obtained if contraindications are present

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Community-dwelling individuals ≥ 60 years who self-identify as men
Enrollment: 60 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Study recruitment rates (feasibility objective) | 12 months
  The study will be considered feasible if the investigators can recruit 12 participants per site within one year
Study retention rates (feasibility objective) | 12 months
  The study will be considered feasible if ≥ 75 % of the sample completes the 12-month assessment
Adherence to the exercise and nutrition interventions (feasibility objective) | 12 months
  The exercise intervention will be considered feasible if participants complete ≥ 65% of the prescribed number of exercise sessions at the 12-month follow-up. The nutrition intervention will be considered feasible if participants attend 66% of the visits.
Perceived usability and satisfaction of the telehealth platform application (feasibility objective) | 12 months
  Measured using the the System Usability Scale (SUS) where scores range from 0 (very poor) to 100 (excellent). Usability will be deemed to be acceptable if the mean SUS score is above 68 (SUS ≥ 68 = average user experience).

SECONDARY OUTCOMES:
Change of health-related quality of life | 0, 6, and 12 months
  Measured using the multi-dimensional, self-administered EuroQol five-dimension (EQ-5D-3L) questionnaire
Change in social isolation | 0, 6, and 12 months
  Measured using the UCLA 3-Item Loneliness Scale questionnaire
Change in the action planning phase of behaviour | 6 and 12 months
  Measured using the Health Action Process Approach (HAPA) questionnaire
Change in self-efficacy, or confidence, for behaviors related to physical activity and calcium intake | 0, 6, and 12 months
  Measured using the Osteoporosis Self-Efficacy Scale (OSES) questionnaire
Change in fear of falling in community-dwelling older adults | 0, 6, and 12 months
  Measured using the seven-item self-administered Falls Efficacy Scale (FES) questionnaire
Change in physical activity | 0, 6, and 12 months
  Measured using the Physical Activity Scale for the elderly (PASE) questionnaire
Change in total protein intake | 2, 6, and 12 months
  Measured in grams using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Change in total calcium intake | 2, 6, and 12 months
  Measured in mg using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Change in vitamin D intake | 2, 6, and 12 months
  Measured in IU using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Change in functional leg muscle strength | 0 and 12 months
  Measured using the 30-second Chair stand test
Change in gait speed | 0 and 12 months
  Measured using the 10-meter walk test
Change in dynamic balance | 0 and 12 months
  Measured using the four-step square test
Change in balance | 0 and 12 months
  Measured using the Short Form Berg Balance Scale (SF BBS-3P)
Number of falls reported | 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months
  Collected using falls calendar
Healthcare utilization | 0, 6 and 12 months
  Collected using healthcare utilization questionnaire
Reporting of safety outcomes (serious and non-serious adverse events) | 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months
  Collected using Adverse Event Reporting

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Morin, MD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - McMaster University, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No